CLINICAL TRIAL: NCT03106142
Title: Improving Current General Practitioners Care: Feasibility and Effectiveness of a Simple Educational Intervention. Knee Osteoarthritis Care: a Quality Improvement in General Practice
Brief Title: Knee Osteoarthritis Care: A Quality Improvement Intervention in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S58815
Record Dates: First submitted 2016-10-26; First posted 2017-04-10 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: intervention, improvement strategy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Intervention group Control group (usual care)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Academic detailing visit arm (Other): The GPs will receive an academic detailing visit by a medical visitor. GPs will receive information on the conservative evidence-based management of knee osteoarthritis with physiotherapy. The information will be summarized on a flyer for the GPs.
  Interventions: Procedure: Academic detailing visit arm
- control group (No Intervention): The two case vignettes will also be presented to GP who did not received the intervention.

INTERVENTIONS:
Procedure: Academic detailing visit arm — General Practitioners in the intervention group will receive one academic detailing visit. During this visit the GPs will receive information about the importance of physical therapy in the non-surgical management of knee osteoarthritis. The information will be summarized on an information leaflet for the GP.
  Arms: Academic detailing visit arm

SUMMARY:
The aim of this study is to improve the referral rates to physiotherapy of patients with knee osteoarthritis. The intervention consists of one academic detailing visit directed to general practitioners (GPs)

DETAILED DESCRIPTION:
In Belgium, referral rates to physiotherapy of patients with knee osteoarthritis are low. A surveys shows that only 11% of the patients with knee osteoarthritis are referred for physiotherapy in an early stage of the disease process. Referral to physiotherapy is common after arthroplasty for revalidation, but not in early stage of the disease process. The aim of this study is to increase the referral rate for physiotherapy in an early stage of the disease process.

One to three times a year, a large part of Belgian GPs receive an academic detailing visit by an independent medical visitors of Farmaka. Farmaka is a non-profit organization, which is sponsored by the government. Each year, three medical and medication-related themes are developed to provide evidence-based and independent information for primary care management. A visit takes about 20 minutes.

The medical visitors of Farmaka will spend 5 minutes of their standard visit to inform GPs about the evidence-based conservative management of knee osteoarthritis with physiotherapy. The information will focus on the referral of patients with knee osteoarthritis to a physiotherapist in an early stage of the disease. To optimize the effect of the referral to physiotherapists, GPs are asked to specify their prescription by adding a clear therapy description 'exercise therapy with aerobic, muscle strengthening and functional exercises'.

This information will be summarized on a flyer. This flyer will be distributed to the GPs at the end of the academic detailing visit. The flyer gives more extended information about the approach and treatment of knee osteoarthritis. The information and flyer will only be distributed to the intervention group.

For the sample size calculation we want to optimize the referral rate to physiotherapists with 15%.

To detect an absolute difference of 15% in referral rate to physiotherapists we need 100 patients in each group ( with significance level of 5%, 1 on 1 allocation and power of 80%). The control group is composed of GPs, visited by Farmaka, who will not receive the additional information on knee osteoarthritis management.

After 6 months the GPs of the intervention and control group will receive two case vignettes on the management of knee osteoarthritis.

The number of referrals to a physiotherapist of the intervention group and the control group will be compared, as well as the number of specified well-directed prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* active GP setting
* visited by independent medical visitors for academic detailing

Exclusion Criteria:

* not willing to participate
* not visited by independent medical visitors for academic detailing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of referrals to physical therapy of patients with knee osteoarthritis | 6 months after intervention
  2 case vignettes were developed to assess GPs' referral rate

SECONDARY OUTCOMES:
Number of technical investigations ordered by GPs for patients with knee osteoarthritis | 6 months after the intervention
  2 case vignettes were developed to assess GPs' request of technical investigations
Type of pain medication prescribed by GPs for patients with knee osteoarthritis | 6 months after the intervention
  2 case vignettes were developed to assess GPs' medication prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Vankrunkelsven, Professor, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

REFERENCES:
- [Background] Habraken H, Janssens I, Soenen K, van Driel M, Lannoy J, Bogaert M. Pilot study on the feasibility and acceptability of academic detailing in general practice. Eur J Clin Pharmacol. 2003 Jul;59(3):253-60. doi: 10.1007/s00228-003-0602-6. Epub 2003 May 22. PMID 12761604
- [Background] May F, Simpson D, Hart L, Rowett D, Perrier D. Experience with academic detailing services for quality improvement in primary care practice. Qual Saf Health Care. 2009 Jun;18(3):225-31. doi: 10.1136/qshc.2006.021956. PMID 19468007